CLINICAL TRIAL: NCT00003077
Title: Phase I/II Trial of Omega-3 Fatty Acids for Cancer Cachexia
Brief Title: Omega-3 Fatty Acids in Treating Patients With Advanced Cancer Who Have Significant Weight Loss
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Alliance for Clinical Trials in Oncology (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: CALGB-9473; U10CA031946 (NIH); CLB-9473; NCI-P97-0097; CDR0000065766 (Registry Identifier: NCI Physician Data Query)
Record Dates: First submitted 1999-11-01; First posted 2003-10-22 (Estimated); Last update posted 2016-07-13 (Estimated); Status verified 2016-07

CONDITIONS: Leukemia; Lymphoma; Multiple Myeloma and Plasma Cell Neoplasm
MeSH Terms: conditions — Leukemia; Lymphoma; Multiple Myeloma; Neoplasms, Plasma Cell | interventions — Fatty Acids, Omega-3

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Omega-3 fatty acid (Experimental): Patients receive omega-3 fatty acids orally in two equal doses with/after breakfast and lunch for 4 months or until weight loss is observed.
  Dose is escalated in cohorts of two patients, although dose escalation is allowed in individual patients. Patients are evaluated for cachexia response every 2 weeks, and tumor response every 4 weeks for a maximum of 4 months. If no response of cachexia or tumor after a 2 month period, patients will be discontinued from study. Patients will be followed for survival post-treatment.
  Interventions: Dietary Supplement: omega-3 fatty acid

INTERVENTIONS:
Dietary Supplement: omega-3 fatty acid

SUMMARY:
RATIONALE: Omega-3 fatty acids are used by the body for energy and tissue development and may be an effective treatment for patients with advanced cancer who are unable to maintain their body weight.

PURPOSE: Phase I/II trial to study the effectiveness of omega-3 fatty acids in treating patients with advanced cancer who have significant weight loss.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine whether omega-3 fatty acids will reverse weight loss in advanced cancer patients with cachexia.
* Determine the maximum tolerated dose (MTD) of omega-3 fatty acids in these patients (phase I completed 12/1999).
* Determine whether omega-3 fatty acids will result in an antitumor response.

OUTLINE: This is a randomized, stratified, dose escalation study. Patients are stratified by the extent of weight loss (2-5 percent or greater than 5 percent in the past month).

Patients receive omega-3 fatty acids orally in two equal doses with/after breakfast and lunch for 4 months or until weight loss is observed.

Dose is escalated in cohorts of two patients, although dose escalation is allowed in individual patients. The maximum tolerated dose (MTD) is defined as the highest dose level at which no greater than one-third of the patients treated, including escalated patients from a lower dose, experience grade 3 or worse toxicity (phase I completed 12/1999).

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically or cytologically proven advanced cancer not amenable to curative therapy (solid tumors and hematologic malignancies eligible except primary and metastatic brain tumors)
* Cachexia (weight loss at least 2 percent within a one month period)

PATIENT CHARACTERISTICS:

Age:

* 18 and over

Performance Status:

* CALBG 0-2

Life Expectancy:

* At least 2 months

Hematopoietic:

* Granulocytes greater than 1,000/mm3
* Platelet count greater than 75,000/mm3
* Hemoglobin greater than 8 mg/dL

Hepatic:

* AST less than 3 times upper limit of normal (ULN)
* Alkaline phosphatase less than 3 times ULN
* Bilirubin less than 1.5 times ULN

Renal:

* BUN less than 1.5 times ULN
* Creatinine less than 1.5 times ULN

Cardiovascular:

* No congestive heart failure requiring diuretics within less than 6 months
* No uncontrolled or severe cardiovascular disease within less than 6 months
* No myocardial infarction within less than 6 months

Other:

* Not pregnant nor contemplating pregnancy during study
* Negative pregnancy test
* No uncontrolled hypercalcemia
* No metabolic disorders (hyperthyroidism)
* No poorly controlled diabetes
* No peripheral edema or ascites requiring diuretics
* No enteric fistulas, with tracheobronchial fistulas or with aspiration
* No esophageal or bowel obstruction that would preclude eating
* Free T4 within normal range
* No serious medical illness
* No psychosis
* No uncontrolled bacterial, viral, or fungal infections
* No active uncontrolled duodenal ulcers
* Above laboratory values required unless bone marrow, liver, kidney, or splenic involvement by tumor is documented

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* Not specified

Chemotherapy:

* Prior and concurrent chemotherapy allowed

Endocrine therapy:

* No concurrent steroids such as dronabinol or megestrol acetate (except for adrenal failure)

Radiotherapy:

* No prior or concurrent radiotherapy to abdomen or pelvis

Surgery:

* Greater than 3 weeks since major surgery
* Greater than 1 week since minor surgery

Other:

* No concurrent diuretics

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 63 (Actual)
Dates: Start 1995-10; Primary Completion 2004-07 (Actual); Study Completion 2004-11 (Actual)

PRIMARY OUTCOMES:
survival | up to 4 months

CONTACTS AND LOCATIONS:
Overall Officials: C. Patrick Burns, MD, Study Chair — Holden Comprehensive Cancer Center
Locations (5):
- United States (5):
  - CCOP - Christiana Care Health Services, Wilmington, Delaware
  - Holden Comprehensive Cancer Center at The University of Iowa, Iowa City, Iowa
  - North Shore University Hospital, Manhasset, New York
  - New York Presbyterian Hospital - Cornell Campus, New York, New York
  - CCOP - Southeast Cancer Control Consortium, Winston-Salem, North Carolina

REFERENCES:
- [Result] Burns CP, Halabi S, Clamon G, Kaplan E, Hohl RJ, Atkins JN, Schwartz MA, Wagner BA, Paskett E. Phase II study of high-dose fish oil capsules for patients with cancer-related cachexia. Cancer. 2004 Jul 15;101(2):370-8. doi: 10.1002/cncr.20362. PMID 15241836